CLINICAL TRIAL: NCT01356576
Title: Effect of Hemodialysis Membranes on Platelet Count
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Edward Epstein, M.D., Northwell Health
Other Study IDs: 10-039
Record Dates: First submitted 2011-05-13; First posted 2011-05-19 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if there is a drop in platelet count after hemodialysis. Hemodialysis membranes are known to activate complement and cause a drop in platelets and sometimes in white blood cells. The investigators are going to study one of the membranes which is the Fresenius Optiflux® to check if it causes a drop in platelets.

ELIGIBILITY:
Inclusion Criteria:

* Patients on Hemodialysis for >=6 months

Exclusion Criteria:

* Hematological Cancers

  * Myelodysplastic syndromes
  * Baseline thrombocytopenia
  * Acute infections (patients on antibiotics)
  * Patients with Immune thrombocytopenic purpura (ITP)/Thrombotic thrombocytopenic purpura (TTP)
  * HIV
  * Liver disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were being selected from the community where undergoing dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Drop in platelet counts | 90 minutes through hemodialysis and immediately after finishing hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Edwerd Epstein, M.D., Principal Investigator — Staten Island University Hospital
Locations (1):
- Island Rehabilitative Service, Staten Island, New York, United States